CLINICAL TRIAL: NCT04764617
Title: Muscle Phenotyping in Frail Older Patients Having Hip Surgery Following Fracture
Brief Title: Functioning of Elder Muscle; Understanding Recovery
Acronym: FEMUR
Status: Active, not recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham Biomedical Research Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20/LO/0841
Record Dates: First submitted 2021-02-08; First posted 2021-02-21 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Frailty Syndrome
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Skeletal Muscle biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
As people get older, the amount of skeletal muscle in the body can decrease. When the amount of this muscle in the body gets very low, there is an increased risk of falling, and not only is recovery to any injury slower, but more complications can be experienced following surgery, and patients may end up being more dependent on the help of others for meeting daily activities. However, it is not clear whether it is simply the amount of muscle that is in the body that is important for health, or whether it is the ability of muscle to function properly which is important.

This research study is looking at the way muscles of frail older people function; not just how strong they are, but the amount of fats and protein that there are in muscle cells, and how the genes in the muscles are being expressed (genes being a collection of chemical information that carry the instructions for making the proteins a cell will need to function).

We will also investigate whether recovery from hip fracture is impacted by the amount of muscle that there is in the body, and/or the functioning of this muscle.

DETAILED DESCRIPTION:
Sarcopenia is the age-associated loss of skeletal muscle mass, muscle quality and strength, and is a contributive factor to frailty in older individuals. Meta-analyses suggest that individuals with sarcopenia appear to be at greater risk of hospitalisation (all cause), falls and fracture, with hip fracture following a fall being both a serious consequence of sarcopenia, as well as a risk factor for frailty syndrome. The short and longer term outcomes for patients who have a hip fracture following a fall are poor (post-operative complications, increased length of hospital stay, and increased mortality risk, institutionalisation and dependency, respectively), and these are understood to be largely due to the underlying vulnerability (frailty) of the people who sustain hip fractures, with poor recovery being compounded by the reduced muscle strength and low muscle mass common in those who are frail.

As a consequence of research on the physiology of ageing muscles and sarcopenia, increasingly there is the possibility that novel agents (such as anabolic agents) could help to alleviate the frailty state in these patients and hence improve shorter and longer term outcomes. However, before novel interventions can be applied to patients with frailty and sarcopenia, such as those sustaining a hip fracture following a fall, an understanding of how the muscles of these patients are functioning at the cellular level, both in the injured and uninjured state is needed; which metabolic pathways are active and which are inactive, those which are enhanced and those which are impaired, so that treatments that are appropriate for the specific metabolic state of these patients can be selected. In recent years there have been advances in the understanding of the cellular physiology of the muscles of older people. However, few of the research studies carried out to date have analysed muscle collected from individuals who are as frail as the patients who present with hip fractures, or probed the metabolic changes which occur in the muscle following injury in this cohort. Findings from cross-sectional investigations on the healthy older person and prospective studies which try and mimic the muscle wasting seen in sarcopenia (using immobilisation or bed rest protocols) could prove useful in this endeavour. However, it is possible that results from these studies may not be generalizable to those who are frail (who may have other clinical problems and take multiple medications) and it is important that deep phenotyping of muscle from these patients is undertaken to address this knowledge gap.

Across the whole study, including a cohort subset, a range of people with frailty, including those with cognitive impairment will be studied. Those with dementia or severe cognitive impairment tend to be those who are most frail and represent a high proportion of patients admitted with a hip fracture. If such patients are excluded, there is a risk of only observing muscle metabolic and histological changes seen in milder levels of frailty, which may not provide a comprehensive picture of sarcopenia. This is a frequent criticism and limitation of previous studies carried out in this field.

Participants will be older individuals admitted to Nottingham University Hospital (UK) with a fractured hip sustained following a fall. In all participants, a muscle sample will be taken from their injured leg during the surgical repair to their hip, with the option for a muscle biopsy to be taken, whilst in theatre, from their uninjured leg using the Bergstrom technique. These samples will be analysed for intramyocellular lipid content and messenger ribonucleic acid (mRNA) expression of 384 gene targets spanning a number of cellular functions. In the week following surgery, measurements of thigh muscle thickness (Ultrasound imaging) and hand grip strength will be made, and an optional assessment of whole body muscle mass using the D3-creatine method will be offered. After discharge from hospital, patient-related outcomes measures will be obtained from medical notes and Three months after surgery, a set of questionnaires will be sent to the participant or their carer to complete. These will assess current mobility, dependency and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Frailty Score (assessed as part of standard care) ≥ 4
* Fractured hip, sustained following a fall, that requires surgery
* Good understanding of spoken and written English language
* Able to give informed consent, or availability of a legally acceptable surrogate to provide consent

Exclusion Criteria:

* Those who fell and sustained their hip fracture greater than 12 hours prior to hospitalisation.
* Those who have fallen and sustained a hip fracture whilst an in-patient in hospital
* Those who sustained the hip fracture as a result of high impact trauma (e.g. road traffic accident)
* Surgery carried out later than 96 hrs after fall
* Chronic neurological, inflammatory or musculoskeletal disorders which result in muscle wasting, e.g. Multiple sclerosis, muscular dystrophy, rheumatoid arthritis
* Any co-morbidity which precludes hip surgery
* Those with a compromised swallowing reflex which would prevent the participant from taking fluids orally, will be excluded.
* Those taking diabetes medication

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Individuals >65 years who have been admitted to Queens Medical Centre, Nottingham, UK for surgical repair of a hip fracture sustained following a low impact fall.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Skeletal Muscle messenger ribonucleic acid (mRNA) expression (injured leg) | On recruitment
  mRNA expression of 384 gene targets spanning a number of cellular functions, in a vastus lateralis muscle biopsy taken from the injured leg

SECONDARY OUTCOMES:
Skeletal Muscle mRNA expression (un-injured leg) | On recruitment
  mRNA expression of 384 gene targets spanning a number of cellular functions, in a vastus lateralis muscle biopsy taken from the uninjured leg
Intramyocellular lipid density (injured leg) | On recruitment
  Intra-myocellular lipid density in a vastus lateralis muscle biopsy taken from the injured leg
Intramyocellular lipid density (uninjured leg) | On recruitment
  Intra-myocellular lipid density in a vastus lateralis muscle biopsy taken from the uninjured leg
Body weight | on recruitment
  body mass (kg)
Grip Strength | up to 3 days post surgery
  Hand grip strength measured on dominant arm - highest of 3 attempts
Groningen Frailty Indicator (GFI) questionnaire | on recruitment
  Groningen Frailty Indicator Score: minimum value (no frailty) indicated by a score of 0, increasing to a maximum value of 15 (completely disabled). Frailty is indicated by a score ≥4, with lower scores indicating better outcomes
Groningen Frailty Indicator (GFI) questionnaire | 1 week post operative
  Groningen Frailty Indicator Score: minimum value (no frailty) indicated by a score of 0, increasing to a maximum value of 15 (completely disabled). Frailty is indicated by a score ≥4, with lower scores indicating better outcomes
Groningen Frailty Indicator (GFI) questionnaire | 90 days post operative
  Groningen Frailty Indicator Score: minimum value (no frailty) indicated by a score of 0, increasing to a maximum value of 15 (completely disabled). Frailty is indicated by a score ≥4, with lower scores indicating better outcomes
Barthel Index for Activities of Daily Living (BADL) questionnaire | on recruitment
  Barthel Index for Activities of Daily Living score: minimum value (totally independent) indicated by a score of 0, increasing to a maximum value of 60 (totally dependent). Lower scores indicate better outcomes
Barthel Index for Activities of Daily Living (BADL) questionnaire | 1 week post operative
  Barthel Index for Activities of Daily Living score: minimum value (totally independent) indicated by a score of 0, increasing to a maximum value of 60 (totally dependent). Lower scores indicate better outcomes
Barthel Index for Activities of Daily Living (BADL) questionnaire | 90 days post operative
  Barthel Index for Activities of Daily Living score: minimum value (totally independent) indicated by a score of 0, increasing to a maximum value of 60 (totally dependent). Lower scores indicate better outcomes
Rivermead Mobility Index (RMI) Questionnaire | on recruitment
  Rivermead Mobility Index score: minimum value (immobile) indicated by a score of 0, increasing to a maximum value of 15. Higher scores indicate better mobility and better outcomes
Rivermead Mobility Index (RMI) Questionnaire | 1 week post operative
  Rivermead Mobility Index score: minimum value (immobile) indicated by a score of 0, increasing to a maximum value of 15. Higher scores indicate better mobility and better outcomes
Rivermead Mobility Index (RMI) Questionnaire | 90 days post operative
  Rivermead Mobility Index score: minimum value (immobile) indicated by a score of 0, increasing to a maximum value of 15. Higher scores indicate better mobility and better outcomes
EuroQoL health-related quality of life questionnaire (EQ-5D) | 1 week post operative
  EuroQoL health-related quality of life questionnaire score: across each of 5 domains, a minimum value of 1 indicates no problems, increasing to a maximum value of 5 indicating an inability to do a task, or an extreme experience of a sensation. Lower scores indicate better outcomes
EuroQoL health-related quality of life questionnaire (EQ-5D) | 90 days post operative
  EuroQoL health-related quality of life questionnaire score: across each of 5 domains, a minimum value of 1 indicates no problems, increasing to a maximum value of 5 indicating an inability to do a task, or an extreme experience of a sensation. Lower scores indicate better outcomes
Vastus lateralis muscle thickness - injured leg | 3 days post operative
  Vastus lateralis muscle thickness measured at the midpoint using ultrasonography
Vastus lateralis muscle thickness - uninjured leg | 3 days post operative
  Vastus lateralis muscle thickness measured at the midpoint using ultrasonography
Whole body muscle mass | 3 days post operative
  whole body muscle mass assessed using the D3-Creatine method
Clinical outcomes; surgical complications | from date of surgery to date of discharge from hospital; up to 90-days after hip surgery
  occurrence of surgical complications audited from patient notes prior to discharge
Clinical outcomes; adverse events during period of hospitalisation | from date of recruitment to date of discharge from hospital; up to 90-days post operative.
  occurrence of adverse events collected throughout period of hospitalisation
Clinical outcomes; length of stay | at discharge from hospital; up to 90 days post hip surgery
  Length of hospitalisation period audited from patient notes prior to discharge
Clinical outcomes; discharge location | at discharge from hospital; up to 90 days post hip surgery
  discharge location audited from patient notes prior to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Ben Ollivere, MBBS, Principal Investigator — University of Nottingham
Locations (1):
- Queens Medical Centre; Department of Orthopaedics, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
gene expression data will be made available in a open access data depository after publication.